CLINICAL TRIAL: NCT03181438
Title: Efficacy of Ultrasound-guided Transverse Abdominal Plane Block for Analgesia in Renal Transplantation
Brief Title: Efficacy Transverse Abdominal Plane (TAP) Block Renal Transplant Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Henrique Cunha Ferraro, Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAP Block Renal Transplant
Record Dates: First submitted 2017-06-03; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Renal Insufficiency, Chronic; Acute Pain; Kidney Transplantation; Anesthesia, Conduction
Keywords: Renal Transplantation; Acute pain; Regional Anesthesia; TAP Block
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP Block (Experimental): The TAP block will be performed under general anesthesia, according to the technique described below:
  * The patient will be placed supine with the abdomen exposed between the iliac crest and the costal margin
  * After skin antisepsis, a high-frequency ultrasound transducer will be placed transversely across the anterior axillary line above the iliac crest
  * In this region, the abdominal musculature (external oblique, internal oblique and transverse abdomen) is identified, and the transverse abdominal plane of the abdomen
  * The needle (BD-A-50mm) will be inserted in the technique "in plane" to the region of the transverse plane of the abdomen, where the solution will be administered.
  * In this group, will be administered 20 mL of 0.375% ropivacaine
  Interventions: Procedure: TAP Block
- Saline Group (Sham Comparator): The block will be performed under general anesthesia, according to the technique described below:
  * The patient will be placed supine with the abdomen exposed between the iliac crest and the costal margin
  * After skin antisepsis, a high-frequency ultrasound transducer will be placed transversely across the anterior axillary line above the iliac crest
  * In this region, the abdominal musculature (external oblique, internal oblique and transverse abdomen) is identified, and the transverse abdominal plane of the abdomen
  * The needle (BD-A-50mm) will be inserted in the technique "in plane" to the region of the transverse plane of the abdomen, where the solution will be administered.
  * In this group, will be administered 20 mL of Saline
  Interventions: Procedure: Saline Group

INTERVENTIONS:
Procedure: TAP Block — It will be performed a ultrasound-guided transverse abdominal plane block with 20 ml of 0.375% of ropivacaine for patients submitted to renal transplantation
  Arms: TAP Block
Procedure: Saline Group — t will be performed a ultrasound-guided transverse abdominal plane block with 2o mL of saline for patients submitted to renal transplantation
  Arms: Saline Group

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of transverse abdominal plane block in patients undergoing renal transplant surgery.Adult renal transplant recipients will be prospectively randomized to receive a standard general anesthetic technique supplemented with ropivacaine 0.375% 20 mL TAP block or sham block with 20 mL 0.9% saline. Both groups will receive patient-controlled morphine analgesia. Patient assessment will occur in the postanesthetic care unit and at 1, 2, 4, 6, 12, and 24 hours. The primary outcome is total morphine consumption in the first 24 hours after renal transplantation. Other outcomes asses include pain scores, presence of nausea or vomiting, excessive sedation, and respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* end-stage renal disease undergoing cadaveric renal transplantation

Exclusion Criteria:

* Contraindications to the use of morphine
* Contraindications to the use ropivacaine
* Peripheral neuropathy
* Inability to use a Patient Control Analgesia device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-06-03 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Morphine Consumption | 24 hours post-operative
  Patient Control Analgesia: morphine sulfate 2 mg IV every 5 minutes until visual analog scale pain score (0 = no pain, 10 = worst possible pain) is 3 or less, and continued at the following settings for a 24-hour period: 1 mg bolus, 7-minute lockout, and 30 mg maximum 4-hourly dose.

SECONDARY OUTCOMES:
Pain Score | 24 hours post-operative
  Visual analogue score (VAS) at rest and movement

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo HC Ferraro, Professor, Principal Investigator — Federal University of São Paulo
Locations (1):
- Hospital do Rim e Hipertensao, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu CL, Raja SN. Treatment of acute postoperative pain. Lancet. 2011 Jun 25;377(9784):2215-25. doi: 10.1016/S0140-6736(11)60245-6. PMID 21704871
- [Result] Dean M. Opioids in renal failure and dialysis patients. J Pain Symptom Manage. 2004 Nov;28(5):497-504. doi: 10.1016/j.jpainsymman.2004.02.021. PMID 15504625
- [Result] Finnerty O, Carney J, McDonnell JG. Trunk blocks for abdominal surgery. Anaesthesia. 2010 Apr;65 Suppl 1:76-83. doi: 10.1111/j.1365-2044.2009.06203.x. PMID 20377549
- [Result] McDonnell JG, O'Donnell BD, Farrell T, Gough N, Tuite D, Power C, Laffey JG. Transversus abdominis plane block: a cadaveric and radiological evaluation. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):399-404. doi: 10.1016/j.rapm.2007.03.011. PMID 17961838
- [Result] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Result] Warman P, Nicholls B. Ultrasound-guided nerve blocks: efficacy and safety. Best Pract Res Clin Anaesthesiol. 2009 Sep;23(3):313-26. doi: 10.1016/j.bpa.2009.02.004. PMID 19862890
- [Result] Niraj G, Searle A, Mathews M, Misra V, Baban M, Kiani S, Wong M. Analgesic efficacy of ultrasound-guided transversus abdominis plane block in patients undergoing open appendicectomy. Br J Anaesth. 2009 Oct;103(4):601-5. doi: 10.1093/bja/aep175. Epub 2009 Jun 26. PMID 19561014
- [Result] Mukhtar K, Khattak I. Transversus abdominis plane block for renal transplant recipients. Br J Anaesth. 2010 May;104(5):663-4. doi: 10.1093/bja/aeq077. No abstract available. PMID 20400617